CLINICAL TRIAL: NCT03031938
Title: A PROTOCOL TO MONITOR FROM BIRTH TO AGE 15 MONTHS THE NEUROLOGICAL DEVELOPMENT OF INFANTS WITH EXPOSURE IN-UTERO IN TANEZUMAB CLINICAL STUDIES AT ALL INVESTIGATIONAL SITES
Brief Title: Protocol to Monitor the Neurological Development of Infants With Exposure in Utero From Birth to 15 Months in Tanezumab Clinical Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A4091065; 2013-002548-10 (EudraCT Number); INFANT SAFETY FOLLOW-UP #2 (Other: Alias Study Number); NEONATAL MONITORING STUDY #2 (Other: Alias Study Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis; Cancer Pain; Recurrent Low Back Pain
Keywords: Exposure in utero in tanezumab program
MeSH Terms: conditions — Osteoarthritis; Cancer Pain; Low Back Pain | interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Other): Long term observational study of subjects from tanezumab parent study
  Interventions: Drug: Investigational medical product (IMP) administered in parent study

INTERVENTIONS:
Drug: Investigational medical product (IMP) administered in parent study — IMP as administered in parent study. IMP would have been either placebo, tanezumab, celecoxib, naproxen, diclofenac, administered in parent study

SUMMARY:
A4091065 is a multicenter, prospective, cohort study with enhance physical an neurodevelopmental surveillance to characterize the outcomes related to the development of infants up to the age of 15 months who were potentially exposed to tanezumab, placebo or comparator via maternal exposure or in utero in any tanezumb study.

DETAILED DESCRIPTION:
A4091065 is a long term observational follow up study of subjects from tanezumab interventional studies A4091056, A4091057, A4091058, A4091059, A4091061 or A4091063

ELIGIBILITY:
Inclusion Criteria:

* Subject is an infant born to a mother who was exposed to study drug on a tanezumab clinical study.
* The infant's mother (who was the tanezumab clinical study participant) must review, agree and sign an informed consent document explaining the details of the perinatal and post natal follow up. Where local regulations mandate, the male parent would also review and sign the informed consent.
* Parents or legal guardian must be willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

* There are no exclusion criteria for participating in this study.

Ages: 0 Years to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - USC Keck School of Medicine, Los Angeles, California
  - Gulfcoast Research Institute, Sarasota, Florida
  - Kennedy and White Orthopaedic Center, Sarasota, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Lafayette Clinical Research Group, Lafayette, Indiana
  - Preferred Pediatrics, Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4091065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants to be enrolled were exposed potentially to tanezumab, placebo or comparator via maternal exposure at conception or in-utero during tanezumab clinical program, in any of the following studies: A4091056 (NCT02697773), A4091057 (NCT02709486), A4091058 (NCT02528188), A4091059 (NCT02528253), A4091061 (NCT02609828) or A4091063 (NCT02725411). Total 4 eligible infants were enrolled. Out of 4, 2 had tanezumab exposure, 2 had comparator (tramadol) exposure and none had placebo exposure.
Pre-assignment Details: Protocol defined visits for vital signs were at age of 0-2, 8 and 15 months. Additional visits to collect vital signs, were defined in 3 month intervals for the first 2 years and then 6 month intervals up till as needed. Neurological examination was planned at age of 0-2, 8 and 15 months. Developmental assessments (BINS, REEL-3) were planned at age of 8 and 15 months. As judged by the investigator neurological examination and developmental assessments could be conducted up to an age 36 months.
Groups:
- Maternal Exposure to Tanezumab: Infants in this reporting arm were those who had potential maternal exposure to tanezumab.
- Maternal Exposure to Tramadol: Infants in this reporting arm were those who had potential maternal exposure to comparator tramadol.
Period: Overall Study
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  Pre-term newborn - gestational age < 37 week | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 0 | 2 | 2
  Race: Black or African American | 1 | 0 | 1
  Race: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Occipital-frontal Head Circumference During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in centimeter (cm) was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: Safety population included all participants who were enrolled into the study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
cm | 38.7 | 38.7 (1.63)

2. Primary Outcome: Occipital-frontal Head Circumference at 8 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in centimeter (cm) was reported.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 47.0 (1.41) | 47.2 (1.44)

3. Primary Outcome: Occipital-frontal Head Circumference at 15 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in centimeter (cm) was reported.
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 49.2 (2.33) | 48.9 (2.69)

4. Primary Outcome: Occipital-frontal Head Circumference During 0 to Less Than or Equal to (<=) 3 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in centimeter (cm) was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
cm | 38.7 | 38.7 (1.63)

5. Primary Outcome: Occipital-frontal Head Circumference During Greater Than (>) 3 to <=6 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in cm was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: Safety population analyzed. "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure. Window period 3 to 6 months was not protocol defined but was an additional window to report data for participants whose initial visit was outside of the protocol defined window of 0-2 months. No participant for reporting arm "Maternal Exposure to Tramadol" had a visit within this window period, hence, for this reporting group no data was collected and reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 44.0 |

6. Primary Outcome: Occipital-frontal Head Circumference During >6 to <=9 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in cm was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 47.0 (1.41) | 47.2 (1.44)

7. Primary Outcome: Occipital-frontal Head Circumference During >15 to <=18 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in cm was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 49.2 (2.33) | 48.9 (2.69)

8. Primary Outcome: Occipital-frontal Head Circumference During >21 to <=24 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in cm was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: Safety population included all participants who were enrolled into the study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Protocol defined mandatory visits were till age of 15 months. No participant visited the site for window period >21 to <=24 months for reporting arm "Maternal Exposure to Tramadol". Hence, for this reporting group no data was collected and reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 49.0 |

9. Primary Outcome: Occipital-frontal Head Circumference During >24 to <=30 Months of Participant's Age
Description: Occipital-frontal head circumference of participants in cm was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: Safety population included all participants who were enrolled into the study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Protocol defined mandatory visits were till age of 15 months. No participant visited the site for window period >24 to <=30 months for reporting arm "Maternal Exposure to Tramadol". Hence, for this reporting group no data was collected and reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 50.5 |

10. Primary Outcome: Body Length During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
cm | 54.6 | 56.5 (1.41)

11. Primary Outcome: Body Length at 8 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: At 8 Months of participant's age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 73.6 (3.45) | 73.7 (1.80)

12. Primary Outcome: Body Length at 15 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: At 15 Months of participant's age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 82.3 (3.95) | 81.3 (0.00)

13. Primary Outcome: Body Length During 0 to <=3 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
cm | 54.6 | 56.5 (1.41)

14. Primary Outcome: Body Length During >3 to <=6 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 72.4 |

15. Primary Outcome: Body Length During >6 to <=9 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 73.6 (3.45) | 73.7 (1.80)

16. Primary Outcome: Body Length During >15 to <=18 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
cm | 82.3 (3.95) | 81.3 (0.00)

17. Primary Outcome: Body Length During >21 to <=24 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 92.5 |

18. Primary Outcome: Body Length During >24 to <=30 Months of Participant's Age
Description: Body length of participants in cm was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
cm | 97.8 |

19. Primary Outcome: Body Weight During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Body weight of participants in kilogram (kg) was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
kg | 3.4 | 5.8 (1.03)

20. Primary Outcome: Body Weight at 8 Months of Participant's Age
Description: Body weight of participants in kilogram (kg) was reported.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
kg | 11.3 (2.50) | 11.6 (0.39)

21. Primary Outcome: Body Weight at 15 Months of Participant's Age
Description: Body weight of participants in kilogram (kg) was reported.
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
kg | 13.6 (2.53) | 13.1 (1.09)

22. Primary Outcome: Body Weight During 0 to <=3 Months of Participant's Age
Description: Body weight of participants in kilogram (kg) was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
kg | 3.4 | 5.8 (1.03)

23. Primary Outcome: Body Weight During >3 to <=6 Months of Participant's Age
Description: Body weight of participants in kg was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
kg | 11.3 |

24. Primary Outcome: Body Weight During >6 to <=9 Months of Participant's Age
Description: Body weight of participants in kg was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
kg | 11.3 (2.50) | 11.6 (0.39)

25. Primary Outcome: Body Weight During >15 to <=18 Months of Participant's Age
Description: Body weight of participants in kg was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
kg | 13.6 (2.53) | 13.1 (1.09)

26. Primary Outcome: Body Weight During >21 to <=24 Months of Participant's Age
Description: Body weight of participants in kg was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
kg | 16.0 |

27. Primary Outcome: Body Weight During >24 to <=30 Months of Participant's Age
Description: Body weight of participants in kg was reported.
Time Frame: Any visit during participants' age above 24 Months up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
kg | 18.4 |

28. Primary Outcome: Systolic and Diastolic Blood Pressure During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in millimeter of mercury (mmHg) was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
mmHg
  Systolic Blood Pressure | 90.0 | NA (NA) — Investigator tried to measure infants blood pressure but could not obtain measurements, hence no data available to report.
  Diastolic Blood Pressure | 60.0 | NA (NA) — Investigator tried to measure infants blood pressure but could not obtain measurements, hence no data available to report.

29. Primary Outcome: Systolic and Diastolic Blood Pressure at 8 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in millimeter of mercury (mmHg) was reported.
Time Frame: At 8 Months of participants' age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 1
mmHg
  Systolic Blood Pressure | 95.5 (19.09) | 82.0
  Diastolic Blood Pressure | 66.0 (8.49) | 40.0

30. Primary Outcome: Systolic and Diastolic Blood Pressure at 15 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in millimeter of mercury (mmHg) was reported.
Time Frame: At 15 Months participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
mmHg
  Systolic Blood Pressure | 94.5 (7.78) | 80.0 (2.83)
  Diastolic Blood Pressure | 58.5 (2.12) | 43.0 (4.24)

31. Primary Outcome: Systolic and Diastolic Blood Pressure During 0 to <=3 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in millimeter of mercury (mmHg) was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
mmHg
  Systolic Blood Pressure | 90.0 | NA (NA) — Investigator tried to measure infants blood pressure but could not obtain measurements, hence no data available to report.
  Diastolic Blood Pressure | 60.0 | NA (NA) — Investigator tried to measure infants blood pressure but could not obtain measurements, hence no data available to report.

32. Primary Outcome: Systolic and Diastolic Blood Pressure During >3 to <=6 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in mmHg was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: Safety population analyzed. Window period 3 to 6 months was not protocol defined but was an additional window to report data for participants whose initial visit was outside of the protocol defined window of 0-2 months. No participant for "Maternal Exposure to Tramadol" had a visit within this window period; for "Maternal Exposure to Tanezumab" site missed to take participants' measurement. Thus, no data was collected and reported for both reporting arms.
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Systolic and Diastolic Blood Pressure During >6 to <=9 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in mmHg was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 1
mmHg
  Systolic Blood Pressure | 95.5 (19.09) | 82.0
  Diastolic Blood Pressure | 66.0 (8.49) | 40.0

34. Primary Outcome: Systolic and Diastolic Blood Pressure During >15 to <=18 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in mmHg was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
mmHg
  Systolic Blood Pressure | 94.5 (7.78) | 80.0 (2.83)
  Diastolic Blood Pressure | 58.5 (2.12) | 43.0 (4.24)

35. Primary Outcome: Systolic and Diastolic Blood Pressure During >21 to <=24 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in mmHg was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
mmHg
  Systolic Blood Pressure | 123.0 |
  Diastolic Blood Pressure | 78.0 |

36. Primary Outcome: Systolic and Diastolic Blood Pressure During >24 to <=30 Months of Participant's Age
Description: Systolic and diastolic blood pressure of participants in mmHg was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
mmHg
  Systolic Blood Pressure | 101.0 |
  Diastolic Blood Pressure | 55.0 |

37. Primary Outcome: Pulse Rate During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: Safety population included all participants who were enrolled into the study. Here, "Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
beats per minute | 124.0 | 144.0 (15.56)

38. Primary Outcome: Pulse Rate at 8 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
beats per minute | 117.0 (15.56) | 121.0 (4.24)

39. Primary Outcome: Pulse Rate at 15 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
beats per minute | 108.5 (20.51) | 116.0 (5.66)

40. Primary Outcome: Pulse Rate During 0 to <=3 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
beats per minute | 124.0 | 144.0 (15.56)

41. Primary Outcome: Pulse Rate During >3 to <=6 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
beats per minute | 128.0 |

42. Primary Outcome: Pulse Rate During >6 to <=9 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
beats per minute | 117.0 (15.56) | 121.0 (4.24)

43. Primary Outcome: Pulse Rate During >15 to <=18 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
beats per minute | 108.5 (20.51) | 116.0 (5.66)

44. Primary Outcome: Pulse Rate During >21 to <=24 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
beats per minute | 118.0 |

45. Primary Outcome: Pulse Rate During >24 to <=30 Months of Participant's Age
Description: Pulse rate of participants in beats per minute was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
beats per minute | 118.0 |

46. Primary Outcome: Temperature During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
degree Celsius | 36.2 | 36.6 (0.08)

47. Primary Outcome: Temperature at 8 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
degree Celsius | 36.3 (0.27) | 36.7 (0.08)

48. Primary Outcome: Temperature at 15 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
degree Celsius | 36.1 (0.47) | 36.5 (0.04)

49. Primary Outcome: Temperature During 0 to <=3 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
degree Celsius | 36.2 | 36.6 (0.08)

50. Primary Outcome: Temperature During >3 to <=6 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
degree Celsius | 36.4 |

51. Primary Outcome: Temperature During >6 to <=9 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
degree Celsius | 36.3 (0.27) | 36.7 (0.08)

52. Primary Outcome: Temperature During >15 to <=18 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
degree Celsius | 36.1 (0.47) | 36.5 (0.04)

53. Primary Outcome: Temperature During >21 to <=24 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
degree Celsius | 36.4 |

54. Primary Outcome: Temperature During >24 to <=30 Months of Participant's Age
Description: Temperature of participants in degree Celsius was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
degree Celsius | 36.3 |

55. Primary Outcome: Respiratory Rate During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: Safety population included all participants who were enrolled into the study. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
breaths per minute | 30.0 | 57.0 (9.90)

56. Primary Outcome: Respiratory Rate at 8 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
breaths per minute | 33.0 (1.41) | 34.0 (2.83)

57. Primary Outcome: Respiratory Rate at 15 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: At 15 Months participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
breaths per minute | 34.0 (14.14) | 27.0 (1.41)

58. Primary Outcome: Respiratory Rate During 0 to <=3 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age from 0 to 3 Months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
breaths per minute | 30.0 | 57.0 (9.90)

59. Primary Outcome: Respiratory Rate During >3 to <=6 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age above 3 Months and up to 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
breaths per minute | 44.0 |

60. Primary Outcome: Respiratory Rate During >6 to <=9 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age above 6 Months and up to 9 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
breaths per minute | 33.0 (1.41) | 34.0 (2.83)

61. Primary Outcome: Respiratory Rate During >15 to <=18 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age above 15 Months and up to 18 Months
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
breaths per minute | 34.0 (14.14) | 27.0 (1.41)

62. Primary Outcome: Respiratory Rate During >21 to <=24 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age above 21 Months and up to 24 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
breaths per minute | 44.0 |

63. Primary Outcome: Respiratory Rate During >24 to <=30 Months of Participant's Age
Description: Respiratory rate of participants in breaths per minute was reported.
Time Frame: Any visit during participants' age above 24 Months and up to 30 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
breaths per minute | 44.0 |

64. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings During 0 to Less Than or Equal to (<=) 2 Months of Participant's Age
Description: Neurologic examination evaluated all cranial nerves except I (smell), IX (taste) and XI (shoulder shrug). Motor examination included evaluation of muscle tone, bulk and movement. Sensory examination included test of temperature and superficial pain (homologous dermatomes using cold tuning fork, neurological examination pin) and deep pain by pressure on achilles tendon. Reflex evaluation included biceps, brachioradialis, patellar, and achilles tendons. Evaluation for persistence of developmental reflexes including Moro reflex, palmar and planter grasp, and tonic neck response was evaluated. Autonomic nervous system evaluation included examination of pupillary reaction, heart rate changes in response to activity, and inquiring about abnormal sweating. Abnormality was determined by the assessor.
Time Frame: Any visit during participants' age from 0 to 2 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

65. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings at 8 Months of Participant's Age
Description: as for outcome 64
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

66. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings at 15 Months of Participant's Age
Description: as for outcome 64
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

67. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings at Follow-up Visit 1 (Month 20 of Participant's Age)
Description: as for outcome 64
Time Frame: Follow-up Visit 1 (At the age of Month 20)
Population: Safety population analyzed. "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure. Protocol defined mandatory visits were till age of 15 months. Investigator upon previous assessment suggested only 1 participant of reporting arm "Maternal Exposure to Tanezumab" to have follow up visit for neurological examination. No participant of reporting arm "Maternal Exposure to Tramadol" was suggested for follow up visit, thus no data reported for this arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

68. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings at Follow-up Visit 2 (Month 26 of Participant's Age)
Description: as for outcome 64
Time Frame: Follow-up Visit 2 (At the age of 26 Months)
Population: as for outcome 67
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

69. Primary Outcome: Bayley Infant Neurodevelopmental Screener (BINS) Total Score at Month 8 of Participant's Age
Description: BINS: a validated instrument designed specifically for a high-risk infant population. It consisted of 11-13 items for different age levels (11 items for participants aged from 3-4 months, 11-15 months, 16-20 months; 13 items for participants aged from 5-6 months, 7-10 months, 21-24 months) to assess cognitive, social, language, gross, and fine motor skills. Each item was scored on a range 0 = non-optimal performance to 1 = optimal performance; BINS total score was sum of scores of each item and it ranged for 11 items from 0 (non-optimal performance) to 11 (optimum performance) and for 13 items from 0 (non-optimal performance) to 13 (optimum performance), higher score indicated better performance.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
units on a scale | NA (NA) — Summarized data was not available, individual BINS total score for 2 participants were 13 and 11 respectively. | NA (NA) — Summarized data was not available, individual BINS total score for 2 participants were 11 and 9 respectively.

70. Primary Outcome: Bayley Infant Neurodevelopmental Screener (BINS) Total Score at Month 15 of Participant's Age
Description: as for outcome 69
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
units on a scale | NA (NA) — Summarized data was not available, individual BINS total score for 2 participants were 11 and 7 respectively. | NA (NA) — Summarized data was not available, individual BINS total score for 2 participants were 11 and 10 respectively.

71. Primary Outcome: Bayley Infant Neurodevelopmental Screener (BINS) Total Score at Follow-up Visit 1 (Month 20 of Participant's Age)
Description: as for outcome 69
Time Frame: Follow-up Visit 1 (At the age of Month 20)
Population: Safety population analyzed. "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure. Protocol defined mandatory visits were till age of 15 months. Investigator upon previous assessment suggested only 1 participant of reporting arm "Maternal Exposure to Tanezumab" to have follow up visit for BINS assessment. No participant of reporting arm "Maternal Exposure to Tramadol" was suggested for follow up visit, thus no data reported for this arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
units on a scale | 7 |

72. Primary Outcome: Bayley Infant Neurodevelopmental Screener (BINS) Total Score at Follow-up Visit 2 (Month 26 of Participant's Age)
Description: BINS: a validated instrument designed specifically for a high-risk infant population. It consisted of 11-13 items for different age levels (11 items for participants aged from 3-4 months, 11-15 months, 16-20 months; 13 items for participants aged from 5-6 months, 7-10 months, 21-24 months) to assess cognitive, social, language, gross, and fine motor skills. Each item was scored on a range 0 = non-optimal performance to 1 = optimal performance; BINS total score was sum of scores of each item and it ranged for 11 items from 0 (non-optimal performance) to 11 (optimum performance) and for 13 items from 0 (non-optimal performance) to 13 (optimum performance), higher score indicated better performance. Data collected at age of 26 months used 24 months' age items.
Time Frame: Follow-up Visit 2 (At the age of Month 26)
Population: as for outcome 71
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
units on a scale | 6 |

73. Primary Outcome: Bzoch-League Receptive Expressive Emergent Language Test 3rd Edition (REEL-3) Language Ability Score at Month 8 of Participant's Age
Description: REEL-3, was designed to identify infants and toddlers who had language impairments or who had other disabilities that affect language development. Caregiver answered interview questionnaire by pediatrician, pediatric neurologist or clinical psychologist for receptive language and expressive language subtests. Each of these 2 sub tests had 66 questions with answer of 'yes = 1' or 'no = 0'. Sum of receptive and expressive language subtests answers was used to calculate REEL-3 language ability total score, with following ranges: <70 (very poor), 70-79 (poor), 80-89 (below average), 90-110 (average), 111-120 (above average), 121-130 (superior), and >130 (very superior). Higher scores indicated better language ability.
Time Frame: At 8 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
units on a scale | NA (NA) — Summarized data was not available, individual REEL-3 language ability total score for 2 participants were 95 and 91 respectively. | NA (NA) — Summarized data was not available, individual REEL-3 language ability total score for 2 participants were 97 and 93 respectively.

74. Primary Outcome: Bzoch-League Receptive Expressive Emergent Language Test 3rd Edition (REEL-3) Language Ability Score at Month 15 of Participant's Age
Description: as for outcome 73
Time Frame: At 15 Months of participants' age
Population: Safety population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 2 | 2
units on a scale | NA (NA) — Summarized data was not available, individual REEL-3 language ability total score for 2 participants were 86 and 89 respectively. | NA (NA) — Summarized data was not available, individual REEL-3 language ability total score for 2 participants were 99 and 97 respectively.

75. Primary Outcome: Bzoch-League Receptive Expressive Emergent Language Test 3rd Edition (REEL-3) Language Ability Score at Follow-up Visit 1 (Month 20 of Participant's Age)
Description: as for outcome 73
Time Frame: Follow-up Visit 1 (At the age of Month 20)
Population: Safety population analyzed. "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure. Protocol defined mandatory visits were till age of 15 months. Investigator upon previous assessment suggested only 1 participant of reporting arm "Maternal Exposure to Tanezumab" to have follow up visit for REEL-3 assessment. No participant of reporting arm "Maternal Exposure to Tramadol" was suggested for follow up visit, thus no data reported for this arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
units on a scale | 88 |

76. Primary Outcome: Bzoch-League Receptive Expressive Emergent Language Test 3rd Edition (REEL-3) Language Ability Score at Follow-up Visit 2 (Month 26 of Participant's Age)
Description: as for outcome 73
Time Frame: Follow-up Visit 2 (At the age of Month 26)
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
Number analyzed (Participants) | 1 | 0
units on a scale | 92 |

ADVERSE EVENTS:
Time Frame: From the participants' age of 0 month to maximum of 36 months
Description: Same event may appear as both adverse event (AE) and serious adverse event (SAE). An event may be categorized as serious in 1 participant and non-serious in other, or participant may experience both SAE and non-SAE.
Arm/Group | Maternal Exposure to Tanezumab | Maternal Exposure to Tramadol
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Exposure to Tanezumab (N=2) | Maternal Exposure to Tramadol (N=2)
Drowning (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Exposure to Tanezumab (N=2) | Maternal Exposure to Tramadol (N=2)
Speech disorder/ Language development delay (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder developmental / Speech developmental delay (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03031938/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03031938/SAP_001.pdf